CLINICAL TRIAL: NCT04670640
Title: Mechanistic Interventions and Neuroscience of Dissociation
Acronym: MIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Negar Fani, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001840; R01AT011267-01 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Dissociation
Keywords: Trauma; PTSD; Mindfulness; Meditation; Neuroimaging; MRI
MeSH Terms: conditions — Dissociative Disorders; Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Breath Focus (Experimental): Participants receiving the breath focus study intervention.
  Interventions: Behavioral: Breath Focus
- Vibration (Experimental): Participants receiving the vibration study intervention.
  Interventions: Device: Vibration
- Vibration With Breath Focus (Experimental): Participants receiving the vibration with breath focus study intervention.
  Interventions: Device: Vibration; Behavioral: Breath Focus
- Screens Free (Experimental): Participants receiving the screens free study intervention.
  Interventions: Behavioral: No Distractions

INTERVENTIONS:
Device: Vibration — Participants will attend two intervention sessions per week for a total of 8 sessions. Participants will sit in a chair in a sound-proof booth monitored by a researcher in front of a computer screen (which delivers instructions) and will be fitted with psychophysiology leads and a device strapped around the chest. There will be no explicit tasks or direction given in this intervention. Participants will experience smooth slowly varying breath-like vibration on their sternum. They will receive their assigned intervention for approximately 18 minutes.
  Arms: Vibration; Vibration With Breath Focus
Behavioral: Breath Focus — Participants will attend two intervention sessions per week for a total of 8 sessions. Participants will sit in a chair in a sound-proof booth monitored by a researcher in front of a computer screen (which delivers instructions) and will be fitted with psychophysiology leads and a device strapped around the chest. The participant will be asked to focus on their breathing during this intervention. They will receive their assigned intervention for approximately 18 minutes.
  Arms: Breath Focus; Vibration With Breath Focus
Behavioral: No Distractions — Participants will attend two intervention sessions per week for a total of 8 sessions. Participants will sit in a chair in a sound-proof booth monitored by a researcher in front of a computer screen (which delivers instructions) and will be fitted with psychophysiology leads and a device strapped around the chest. Participants will engage in a period of no-screen time; during this time there will be no outside visual or auditory distractions. There will be no explicit tasks or direction given in this intervention. They will receive their assigned intervention for approximately 18 minutes.
  Arms: Screens Free

SUMMARY:
The purpose of this study is to test the neurophysiological mechanisms of an intervention to reduce symptoms of dissociation in traumatized people. The intervention will be tested in dissociative traumatized people at two sites: Emory University and University of Pittsburgh. The researchers are interested in whether neural networks associated with attentional control and interoceptive awareness can be enhanced in this population. The researchers propose to evaluate whether different body-focused and non-body focused interventions can change these mechanisms.

DETAILED DESCRIPTION:
People exposed to chronic trauma face devastating effects to the brain and body. Chronically traumatized people become highly distressed when attending to emotional stimuli, which can lead to feelings of detachment from their bodies and environment. It is difficult to engage highly dissociative traumatized patients in trauma-focused treatment; however, these patients benefit from acquiring basic emotion regulation skills, including present-centeredness and body awareness. Various practices that involve present-centeredness and body awareness (including mindfulness-based interventions) have been shown to demonstrate short-term and long-term improvement in cognition, emotion regulation and clinical symptoms in dissociative people with trauma exposure.

In order to address this issue, the researchers will evaluate the effectiveness of interventions that engage present-centered awareness and/or body focus.

ELIGIBILITY:
Inclusion Criteria:

* experience of at least one Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Criterion A trauma (assessed using the Life Events Checklist)
* a score of 7 or higher on the Multiscale Dissociation Inventory (MDI) depersonalization subscale
* willingness to participate in the study

Exclusion Criteria:

* actively psychotic and cognitively compromised individuals (assessed using the Moderate-severe cognitive impairment screening tool (MoCA) will be excluded
* moderate or more severe substance dependence (assessed with the MINI)
* persons with imminent risk of physical violence to self or others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered Post Traumatic Stress Disorder (PTSD) Scale (CAPS) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The CAPS is a 30-item structured interview that can be used to make current and lifetime diagnosis of post traumatic stress disorder (PTSD) as well as assess PTSD symptoms over the past week. Questions also examine the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization). The identification of an index traumatic event to serves as the basis for symptom inquiry. The full interview takes approximately 45-60 minutes to administer. Items are scored from 0 to 4 where 0 = the symptom is absent and 4 = the symptom is incapacitating. A symptom severity score is obtained by summing items 1-20. Total scores range from 0 to 80 and a higher score indicates more severe PTSD symptoms.
Change in Mini International Neuropsychiatric Interview (MINI) Diagnosis of Psychiatric Disorders | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Mini International Neuropsychiatric Interview (MINI) is a semi-structured interview used for diagnosing psychiatric disorders. The number of participants diagnosed with psychiatric disorders at the study time points will be compared between study arms.
Change in Multiscale Dissociation Inventory (MDI) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The MDI is a 30-item self-report test of dissociative symptomology and measures six different types of dissociative responses: disengagement, depersonalization, derealization, emotional constriction/numbing, memory disturbance, and identity dissociation. Items are scored on a 5-point scale where 1 = never and 5 = very often. Total dissociation scores range from 30 to 150 where higher scores indicate greater symptoms of dissociation.
Change in Kentucky Mindfulness Scale (KIMS) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Kentucky Mindfulness Scale is a 39-item scale that assesses skills related to what one does while practicing mindfulness. Items are rated on a 5 point Likert scale ranging from 1 (never or very rarely true) to 5 (almost always or always true). Items reflect either direct descriptions of the mindfulness skills, or they describe the absence of that skill and are reverse scored. Total scores range from 39 to 195 and higher scores reflect more mindfulness.
Change in Multidimensional Assessment of Interoceptive Awareness (MAIA) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  This is a clinical measure that assesses various aspects of interoception, including ability to attend to body sensations, regulate distress by attending to body sensations, and experiencing body sensations as safe and trustworthy. The instrument includes 32 items and which are scored from 0 to 5, where 0 = never and 5 = always. Total scores range from 0 to 160 and higher scores indicate greater awareness of body sensations.
Change in Attentional Control Scale (ACS) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  This is a 20-item self-report measure that assesses attentional control a 4-point Likert scale, where 1 = almost never and 4 = always. Total scores range from 20 to 80 and higher scores indicate greater difficulty with attentional control.
Change in Difficulties in Emotion Regulation Scale (DERS) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The DERS is a 36 item instrument that measures emotional dysregulation symptoms. Responses are given on a 5-point scale where 1 = almost never and 5 = almost always. The DERS scales include 1) nonacceptance of emotional responses, 2) difficulty engaging in goal-directed behavior, 3) difficulties with impulse control, 4) limited emotional awareness, 5) limited access to emotion regulation strategies, and 6) lack of emotional clarity. Total scores range from 36 to 180 and higher scores suggest greater problems with emotion regulation.
Change in PTSD Symptom Checklist (PCL-5) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The PCL-5 is a 20-item self-report measure that assess the DSM-V symptoms of PTSD. Responses are given on a scale from 0 to 4 where 0 = not at all and 4 = extremely. Total scores range from 0 to 80 where higher scores indicate increased symptoms of PTSD.
Change in Change in Life Events Checklist Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Life Events Checklist includes 21 items asking respondents if they have been exposed to stressful events in the last 3 to 4 weeks. Participants are also able to list stressful events or experiences that are not specifically listed. Responses are coded as 5 = happened to me, 4 = witnessed it, 3 = learned about it, 2 = part of my job, 1 = not sure, and 0 = does not apply. A total score or composite score is not calculated for the Life Events Checklist, rather this instrument is used to identify if the respondent has experienced traumatic situations.
Change in Sense of Agency Rating Scale (SOARS) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The SOARS is a 10-item self-report measure that assess the sense of control one has over their body. Responses are given on a 7-point Likert scale where 1 = strongly disagree and 7 = strongly agree. Total scores range from 10 to 70 where lower scores indicate greater sense of agency.
Change in Primary Care PTSD Screen (PC-PTSD-5) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The PC-PTSD-5 is a 5-item instrument is used to identify persons with probable PTSD. Participants reporting that they have experienced a traumatic event are asked if they have had certain symptoms of PTSD in the past month. Responses are scored as no = 0 and yes = 1. Total scores range from 0 to 5 with higher scores indicating increased symptoms of PTSD.
Change in Scale of Body Connection (SBC) Body Awareness Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Scale of Body Connection instrument has 20 items assessing the dimensions of Body Awareness and Bodily Dissociation. Items are scored on a 5-point scale where 0 = not at all and 4 = all of the time. The body awareness dimension has 12 items and the body awareness score is the average of responses to these items. Higher scores indicate greater bodily awareness.
Change in Scale of Body Connection (SBC) Bodily Dissociation Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Scale of Body Connection instrument has 20 items assessing the dimensions of Body Awareness and Bodily Dissociation. Items are scored on a 5-point scale where 0 = not at all and 4 = all of the time. The bodily dissociation dimension has 8 items and the bodily dissociation score is the average of responses to these items. Higher scores indicate greater bodily dissociation.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Alcohol Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime alcohol use with up to 7 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 13 where higher scores indicate greater lifetime use of alcohol.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Alcohol 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses alcohol use in the last 30 days with up to 4 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 13 where higher scores indicate greater use of alcohol in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Tobacco Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime tobacco use with up to 8 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 13 where higher scores indicate greater lifetime use of tobacco.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Tobacco 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses tobacco use in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater use of tobacco in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Cocaine Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime cocaine use with up to 7 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 16 where higher scores indicate greater lifetime use of cocaine.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Cocaine 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses cocaine use in the last 30 days with up to 4 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 13 where higher scores indicate greater use of cocaine in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Heroin Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime heroin use with up to 8 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 13 where higher scores indicate greater lifetime use of heroin.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Heroin 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses heroin use in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 13 where higher scores indicate greater use of heroin in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Illicit Opiate Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime illicit use of prescription opiates with up to 8 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater lifetime illicit use of prescription opiates.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Illicit Opiates 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses illicit use of prescription opiates in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 11 where higher scores indicate greater illicit use of prescription opiates in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Marijuana/Cannabis Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime marijuana/cannabis use with up to 7 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 14 where higher scores indicate greater lifetime use of marijuana/cannabis.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Marijuana/Cannabis 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses marijuana/cannabis use in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater use of marijuana/cannabis in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Amphetamine/Methamphetamine Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime amphetamine/methamphetamine use with up to 7 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater lifetime use of amphetamine/methamphetamine.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Amphetamine/Methamphetamine 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses marijuana/cannabis use in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 11 where higher scores indicate greater use of amphetamine/methamphetamine in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Illicit Benzodiazepines Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime illicit use of benzodiazepines with up to 7 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater lifetime illicit use of benzodiazepines.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Illicit Benzodiazepines 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses illicit use of benzodiazepines in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 11 where higher scores indicate greater illicit use of benzodiazepines in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Benzodiazepines Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime use of healthcare provider prescribed benzodiazepines with up to 7 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater lifetime use of healthcare provider prescribed benzodiazepines.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Benzodiazepines 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses use of healthcare provider prescribed benzodiazepines in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 11 where higher scores indicate greater use of healthcare provider prescribed benzodiazepines in the past 30 days.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Barbiturates Lifetime Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses lifetime use of barbiturates with up to 8 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 12 where higher scores indicate greater lifetime use of barbiturates.
Change in Kreek-McHugh-Schluger-Kellogg Scale (KMSK) Barbiturates 30 Day Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The KMSK assesses use of barbiturates in the last 30 days with up to 5 items. Three of the items are scored quantitatively on varying scales. Total scores range from 0 to 11 where higher scores indicate greater use of barbiturates in the past 30 days.
Change in Patient-Reported Outcomes Measurement Information System - Depression (PROMIS-D) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The PROMIS-D instrument assesses depression with 9 items asking respondents if they have experienced certain symptoms of depression in the past 7 days. Responses are given on a 5-point scale. Total scores are transformed to a t-score with a mean of 50 and standard deviation of 10. Scores above 50 indicate increased depressive symptoms compared to the reference population.
Change in International Trauma Questionnaire Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The International Trauma Questionnaire is an instrument used to diagnose PTSD or complex PTSD (CPTSD) with 18 items (9 items for each of the PTSD and CPTSD subscales). Responses are given on a 5-point scale where 0 = not at all and 4 = extremely. Dimensional scores for PTSD and the Disturbances in Self-Organization (DSO) cluster of the CPTSD subscale can be calculated by summing six items from their respective subscales. Total scores for each subscale range from 0 to 24 with higher values indicating increased problems following experiencing a traumatic event.
Change in Childhood Trauma Questionnaire (CTQ) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Childhood Trauma Questionnaire (CTO) has 28 items asking respondents if they experienced situations of trauma as a child or teenager. Responses are given on a 5-point scale where 1= never true and 5 = always true. There are subscales for sexual abuse, physical abuse, emotional abuse, emotional neglect, and physical neglect, and a total trauma score is calculated. Total scores range from 28 to 140 where higher scores indicate more severe trauma.
Change in Motivation and Pleasure Scale Self-Report (MAP-SR) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The MAP-SR is an 18-item questionnaire assessing the degree of pleasure experienced with social, work or recreational, and family situations and the amount of motivation to engage in activities. Responses are given on a 5-point scale where 0 = no pleasure or no motivation and 4 = extreme pleasure or motivation. Total scores range from 0 to 72. Scoring for certain items is reversed so that higher scores indicate increased pleasure and motivation.
Change in Ruminative Responses Scale Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Ruminative Responses Scale is a 22-item instrument assessing different things that people do when they feel depressed. Responses are given on a 4-point scale where 1 = almost never and 4 = almost always. Total scores range from 22 to 88 and higher scores indicate greater rumination on depressive symptoms, potentially prolonging depressive episodes.
Change in Everyday Discrimination Scale (EDS) Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The original Everyday Discrimination Scale includes 9 items asking respondents how often they experience certain situations of discrimination. Responses are given on a 6-point scale where 1 = never and 6 = almost everyday. Total scores range from 9 to 54 where higher scores indicate experiencing increased discrimination.
Change in Experiences of Discrimination (EOD) Scale Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Experiences of Discrimination Questionnaire is an 11-item instrument assessing experiences of discrimination because of race, ethnicity, or color. Respondents indicate if they have or have not experienced 9 situations of discrimination (no = 0 and yes = 1), and then there are two questions about how often respondents feel that discrimination occurs that are score as 1 = never and 4 = often. Total scores range from 2 to 17 where higher scores indicate greater experiences of discrimination.
Change in Epworth Sleepiness Scale Score | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Epworth Sleepiness Scale is an 8-item instrument assessing level of daytime sleepiness. Responses are given on a 4-point scale where 0 = would never doze and 3 = high chance of dozing. Total scores range from 0 to 24, where scores between 0 and 10 are considered normal and scores above 16 are indicative of high levels of excessive daytime sleepiness.
Change in Penn Computerized Neuropsychological Battery (Penn CNP) Performance | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  This is a computerized neuropsychological assessment that is designed to examine different domains of cognitive functioning. The executive functioning and memory components of this battery (which include measures of sustained attention and working memory) will be administered, which take approximately 30 minutes to complete.
Change in State Scale of Dissociation (SSD) Score | Baseline to Week 6 (before and after each study visit)
  The SSD is a 56-item self-report measure that assess present state dissociative symptoms. The SSD seven subscales are derealization, depersonalization, identity confusion, identity alteration, conversion, amnesia, and hypermnesia. Responses are given on a 10-point scale where 0 = not at all, and 9 = very much so. A total score is calculated as the mean of all survey items. Total scores range from 0 to 9 where higher scores indicate greater dissociation. This will be administered prior to and after each intervention appointment and MRI visit.
Change in Affective Number Stroop (ANS) Task Performance | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  During the ANS task, participants are instructed to rapidly identify the number of numbers in a given display while ignoring evocative distractor images (trauma-relevant scenes). In these trials, the number of numbers presented is either consistent or inconsistent with the actual number displayed, such that there are both congruent and incongruent trials. The participants will be presented with positive and neutral pictures in addition to the negative trauma-relevant images. The task will be completed in the MRI scanner during both the pre- and post-treatment sessions. This task is meant to evoke the attentional problems that many Grady Trauma Project participants encounter while performing daily tasks by engaging attentional control resources and including images that are relevant to participants' traumas.
Change in Stroop Color and Word Test (SCWT) Time | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  During the Stroop Color and Word Test, lists of color words printed in black ink, printed in ink the color of the word, and printed in ink in a color that does not match the word. Participants are asked to read the words in the first two conditions but to then state the color of the ink rather than the word during the inconsistent color condition. The SCWT shows that people take longer to name the color of the ink that color-words are written in when the ink color does not match the word than when they match. The time it takes to complete condition where the ink color does not match the word will be assessed in seconds.
Change in Number Stroop Test Time | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  The Counting Stroop is a validated Stroop task variant. In this task, participants report the number of words (one to four) appearing on the screen, regardless of word meaning, by pressing a button. Neutral-word control trials contain single semantic category common animals (i.e. dog written three times) while interference trials contain number words that are incongruent with the correct response (i.e. 'two' written four times). The time it takes to say the number of words will be assessed in seconds.
Change in Pittsburgh EEG Accessible Calibration Environment (PEACE) Performance | Baseline, Week 6 (post-intervention), 3 Months Post-intervention, 6 Months Post-intervention
  This 6-minute task consists of multiple common cognitive and affective operations including open and closed eyes resting state, passive viewing of affective images, rumination, counting backwards, and finger movement. It allows derivation of physiological profiles for use in signal classification on the other tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Negar Fani, PhD, Principal Investigator — Emory University; Greg Siegle, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Grady Hospital, Atlanta, Georgia
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical and neuroimaging data will be shared. Data will be uploaded continuously to a public repository for clinical trials (e.g., NDAR) as specified by the program official.
Supporting Information: SAP
Time Frame: Data will be available for sharing prior to publication of the study results.
Access Criteria: Data will be made available to the public by inclusion in public repository. Once data are included in a public repository they can be accessed by the public for any reason without contacting the study Principal Investigators.